CLINICAL TRIAL: NCT02588326
Title: Evaluation of the Sensitivity of Pharmacokinetics to Differences in the Particle Size Distribution of Two Different Formulations of a Locally-acting Mometasone Furoate Suspension-based Nasal Spray
Brief Title: Sensitivity of Pharmacokinetics to Differences in Particle Size Distribution of Suspension-based Nasal Sprays
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRB201500381 - F; HHSF223201310220C (Other Grant/Funding Number: US FOOD AND DRUG ADMN); OCR19758 (Other: UF OnCore)
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Hypersensitivity
Keywords: Bioequivalence; Suspension nasal spray; Mometasone furoate; Pharmacokinetics; Particle size distribution
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MFF 1, then MFF 2 (Active Comparator): Mometasone furoate drug formulation (MFF) 1 will be administered by suspension-based nasal spray. After a wash out period then Mometasone furoate drug formulation (MFF) 2 will be administered by suspension-based nasal spray. All formulations will be a 200 mcg single dose.
  Interventions: Drug: Mometasone furoate drug formulation (MFF) 1; Drug: Mometasone furoate drug formulation (MFF) 2
- MFF 2, then MFF 1 (Active Comparator): Mometasone furoate drug formulation (MFF) 2 will be administered by suspension-based nasal spray. After a wash out period then Mometasone furoate drug formulation (MFF) 1 will be administered by suspension-based nasal spray. All formulations will be a 200 mcg single dose.
  Interventions: Drug: Mometasone furoate drug formulation (MFF) 1; Drug: Mometasone furoate drug formulation (MFF) 2

INTERVENTIONS:
Drug: Mometasone furoate drug formulation (MFF) 1 — Mometasone furoate drug formulation (MFF) 1 will be administered by suspension-based nasal spray.
  Other Names: Nasonex re-engineered version
Drug: Mometasone furoate drug formulation (MFF) 2 — Mometasone furoate drug formulation (MFF) 2 will be administered by suspension-based nasal spray.
  Other Names: Nasonex re-engineered version

SUMMARY:
Currently FDA does not accept pharmacokinetic studies to show bioequivalence of locally-acting nasal suspension formulations.

However, bioequivalence is defined as the absence of significant differences in pharmacokinetics of therapeutically equivalent drug products compared to the matching originally invented drug formulation. These there-called "generic drugs" are then interchangeable. Drug companies have to show that their generic version has the same active ingredient, the same label, is intended to be used for the same conditions or diseases and works at the same rate in the body.

The aim of the study is to determine if pharmacokinetics is sensitive to differences in the particle size distribution of two different nasal suspension formulations of mometasone furoate during charcoal block. The result from this study will aid the FDA in finding methods to ensure that generic products are the same as the trade name drugs.

DETAILED DESCRIPTION:
For every subject in this research study the following procedures and scheduling will take place.

During the screening visit the inclusion and exclusion criteria will be reviewed to ensure the subject is appropriate for the study. A physical examination will be performed after the vital sign measurements are obtained. Also, nasal spray application training will be performed and tolerability to charcoal block will be determined.

Screening tests will be performed within 30 days of study visit 1 and no later than 2 days before study visit 1. There will be 2 study visits in addition to the screening visit, a minimum period of 7 days should lapse between the subsequent study visits but no more than 3 weeks. The total study duration for each subject will be about 4-7 weeks.

Blood sample collection

Blood samples will be drawn by inserting an indwelling catheter for blood sample collection. Blood samples will be taken approximately 15 minutes prior to the dosing of the product (pre-dose sample) and at approximately 5, 10, 15, 30, 45, 60 minutes, 1.5, 2, 3, 4, 6, 8, 10, 12 and 14 hours post dosing. At each time point about 10 mL of blood sample will be collected via vacutainer tubes for plasma preparation and storage. At each study visit a total of approximately 160 mL blood will be collected, which makes a total of 320 mL of blood during study visits 1 and 2.

The total amount of blood drawn in this study, including the screening visit, will be 327 ml. Additionally, up to approximately 15 mL of blood may be drawn for medically needed additional assessments to follow up the screening results. Therefore, in total up to approximately 342 mL of blood may be drawn from each subject.

ELIGIBILITY:
Inclusion Criteria

* Healthy male or female subjects aged 18 to 50 years (inclusive).
* Females will be eligible only if they are currently non-lactating and demonstrate a negative urine pregnancy test. Female subjects must be willing to use highly effective methods of contraception throughout the study. A highly effective method of birth control is defined as one which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly e.g. no sexual intercourse, using contraceptive foam AND a condom (double-barrier). [NOTE: for this study, use of hormonal contraception is an exclusion]
* Body mass index (BMI) between 18.5 and 30.0 kg/m2.
* Non-smoker for at least 12 months prior to study screening and a maximum smoking history of less than ten-pack years (i.e. the equivalent of one-pack per day for ten years).
* Free of significant abnormal findings as determined by medical history, physical examination, vital signs, and laboratory tests (including serum cortisol at screening), complete blood count (CBC) with differential , urinalysis and basic metabolic panel.
* Ability to read, comprehend and sign the informed consent form.
* Ability and willingness to comply with all study procedures, discontinue and/or withhold medications as specified in the protocol, and attend scheduled study visits.
* No history of major respiratory disease (such as cystic fibrosis or COPD).
* Able to demonstrate correct nasal spray technique at screening.

Exclusion Criteria

* Any history and/or conditions that might interfere with drug absorption, distribution, metabolism or excretion of MF, e.g., preexisting lung and liver disease.
* Known or suspected sensitivity or allergic reaction to MF, or related compounds in that class, or one of the excipients, or to activated charcoal.
* Known or suspected sensitivity to benzalkonium chloride or to products containing this salt.
* Having a history and/or currently having the medical condition in the opinion of medically accountable investigator and hence taking any medication for the following (including but not limited to):

  * Significant cardiac, dermatologic, gastrointestinal, hepatic, renal, hematological, neurological and psychiatric disease (determined by physical exam, CBC with differential, urinalysis, basic metabolic panel and medical history).
  * Presence of glaucoma, cataracts, ocular herpes simplex or carcinoma (other than basal cell).
  * Presence of tuberculosis and other respiratory diseases (including but not limited to intermittent or persistent asthma, emphysema and chronic bronchitis); or respiratory infection, common cold, sinusitis or ear infections.
* Based on the medical interview, physical examination or screening investigations, subject is unfit for the study in the opinion of the medically accountable investigator.
* Current use of hormone replacement therapy (HRT), hormonal contraceptives (oral, implants, or IUDs) and/or use corticosteroid within the last 2 month.
* Atrophic rhinitis or rhinitis medicamentosa within the last 60 days.
* Any history of nasal surgery or known clinically relevant abnormalities, such as rhinitis medicamentosa, polyposis, septum deviation with clinical symptoms, recent nasal trauma, or nasal structural abnormalities.
* History of recurrent epistaxis, or any epistaxis requiring medical intervention.
* Known perennial airway allergies or vasomotor rhinitis.
* Known seasonal airway allergies within the last six weeks prior to the start of the study or seasonal airway allergies that likely become acute during the study period. Subjects may be included in the study, if e.g. a mild or unlikely seasonal airway allergy does not interfere with the nasal absorption of mometasone furoate in the opinion of the medically accountable investigator and principal investigator.
* Acute sinusitis within the last six weeks prior to enrollment.
* History of chronic sinus disease or sinusitis within the last year prior to the start of study.
* Use of any systemic, topical, inhaled, or nasal corticosteroid within 30 days prior to enrollment.
* Use of any prescription, over-the-counter, or complementary nasally administered products within 30 days prior to enrollment and for the duration of the study (i.e., corticosteroids, decongestants, antihistamines, saline sprays, sinus washes).
* Use of any topically applied agents to the nasal mucosa (i.e., antibacterial creams, Vaseline) within 30 days of enrollment.
* History of malignancy within the past five years.
* Any concurrent medication or any medication within 2 weeks preceding the start of the study (infrequent intake/use of drugs may be accepted, if judged by the investigator to have no clinical relevance and no influence on study outcome).
* Exposure to any investigational drug within 30 days of enrollment. Exposure to any medication/food that alters the CYP 3A4 activity within last 2 weeks (e.g. any grapefruit products, azole anti-fungals, or rifampin).
* Subjects who have donated 14.85 ounces (450 mL) blood or more within the previous 8 weeks prior to study administration.
* Any history of current drug or alcohol abuse, which would interfere with the subject's completion of the study and with adherence to the protocol.
* Subject reports a regular xanthine consumption of > 5 cups of coffee or black tea per day (or equivalent xanthine consumption per day using other products).
* Subject reports strict dietary habits, which would preclude the subject's acceptance of standardized meals.
* A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, co-investigators, study coordinator, or employee of the participating investigator.
* The subject is a student of the Principal Investigator or co-investigators.
* Lack of willingness to have personal study related data collected, archived and transmitted according to the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of mometasone furoate formulation 1 | 15 min pre-dose and 5, 10, 15, 30, 45, 60 minutes and 1.5, 2, 3, 4, 6, 8, 10, 12 and 14 hours post-dose
Area under the plasma concentration versus time curve (AUC) of mometasone furoate formulation 2 | 15 min pre-dose and 5, 10, 15, 30, 45, 60 minutes and 1.5, 2, 3, 4, 6, 8, 10, 12 and 14 hours post-dose

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of mometasone furoate formulation 1 | 15 min pre-dose and 5, 10, 15, 30, 45, 60 minutes and 1.5, 2, 3, 4, 6, 8, 10, 12 and 14 hours post-dose
Peak Plasma Concentration (Cmax) of mometasone furoate formulation 2 | 15 min pre-dose and 5, 10, 15, 30, 45, 60 minutes and 1.5, 2, 3, 4, 6, 8, 10, 12 and 14 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Jurgen Bulitta, PhD, Principal Investigator — University of Florida jbulitta@cop.ufl.edu
Locations (1):
- Department of Pharmaceutics, University of Florida, Gainesville, Florida, United States